CLINICAL TRIAL: NCT02420587
Title: Phase 2 Study of AMG 208 Evaluating the Tumor Microenvironment in Metastatic Castration-Resistant Prostate Cancer
Brief Title: AMG 208 Tumor Microenvironment in Metastatic Castration Resistant Prostate Cancer (mCRPC)
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2013-1049
Record Dates: First submitted 2015-04-15; First posted 2015-04-20 (Estimated); Last update posted 2015-04-20 (Estimated); Status verified 2015-04

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; Adenocarcinoma of the prostate; Castration resistant prostate cancer metastatic to bone; mCRPC; AMG 208; Questionnaire; Survey
MeSH Terms: conditions — Prostatic Neoplasms | interventions — AMG 208; Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- AMG 208 (Experimental): Dose of AMG 208 is 400 mg by mouth daily given in 6 weeks cycles. Participants receive AMG 208 until radiographic progression of disease and/or unequivocal clinical progression. Questionnaire completion about pain at baseline, Day 22 of Cycle 1, Day 1 of Cycle 2, Day 22 of Cycle 2, every 6 weeks, and at end of study visit.
  Interventions: Drug: AMG 208; Behavioral: Questionnaire

INTERVENTIONS:
Drug: AMG 208 — Dose of AMG 208 is 400 mg by mouth daily given in 6 weeks cycles.
Behavioral: Questionnaire — Questionnaire completion about pain at baseline, Day 22 of Cycle 1, Day 1 of Cycle 2, Day 22 of Cycle 2, every 6 weeks, and at end of study visit.
  Other Names: Survey

SUMMARY:
The goal of this clinical research study is learn how AMG208 may help to control prostate cancer that has spread to the bone. The safety of the drug will also be studied.

DETAILED DESCRIPTION:
Study Drug Administration:

If participant is found to be eligible to take part in this study, they will take capsules of AMG208 by mouth 1 time every day while they are on study.

Participant should fast (not have anything except water) for 2 hours before and 1 hour after they take the AMG208 capsules.

Participant will be asked to keep a diary to help them keep track of when they take each dose of the study drug. Participant should record any missed or vomited doses in the diary. If participant vomits their dose, they should not re-take their dose. Participant should wait until their next scheduled dose. Participant should bring the diary with them to each visit.

Every 6 weeks is considered a cycle. Participant should return all unused study drug and/or empty pill bottles at the end of each cycle.

Study Visits:

On Day 1 of Cycle 1 (+/ - 3 days):

* Blood (about 3-4 tablespoons) will be drawn for biomarker testing.
* Participant will have a bone marrow aspiration and biopsy to check the status of the disease and for biomarker testing. To collect a bone marrow aspirate/biopsy, an area of the hip is numbed with anesthetic, and a small amount of bone marrow and bone is withdrawn through a large needle. Biomarkers are found in the blood/tissue and may be related to participant's reaction to the study drug.

On Day 22 of Cycle 1:

* Participant will have a physical exam.
* Participant will have an EKG. Participant will have 2 more EKGs if the study doctor thinks it is needed.
* Blood (about 3-4 tablespoons) and urine will be collected for routine tests. This blood will also be used to check participant's PSA level, to measure CTCs, and for biomarker testing.
* Participant will fill out the questionnaire about pain.

On Day 1 of Cycles 2 and every 6 weeks after that:

* Participant will have a physical exam.
* Blood (about 3-4 tablespoons) and urine will be collected for routine tests. This blood will also be used to check participant's PSA and testosterone levels.
* Participant will fill out the questionnaire about pain.

On Day 1 of Cycles 2 and 3, and every 12 weeks after that:

* Participant will have a bone scan and a CT or MRI scan of the chest, abdomen, pelvis, and any other area the study doctor thinks is needed to check the status of the disease.
* Participant will have an EKG. Participant will have 2 more EKGs if the study doctor thinks it is needed.
* Blood (about 2-3 tablespoons) will be drawn to check participant's thyroid function, and for CTC and biomarker testing.
* Participant will have either an ECHO or a MUGA scan. (Cycles 2 and 5 only and every 12 weeks after that)

On Day 1 of Cycle 2 participant will have a bone marrow aspiration and biopsy to check the status of the disease.

On Day 22 of Cycle 2:

* Participant will have a physical exam.
* Blood (about 3-4 tablespoons) and urine will be collected for routine tests. This blood will also be used to check participant's PSA level.
* Participant will fill out the questionnaire about pain.

On Day 1 of Cycle 5, participant will have a bone marrow aspiration to check the status of the disease.

Length of Study:

Participant may continue taking the study drug for as long as the doctor thinks it is in their best interest. Participant will no longer be able to take the study drug if the disease gets worse, if intolerable side effects occur, or if they are unable to follow study directions.

Patient's participation on the study will be over after the follow-up visit.

End-of-Study Visit:

If they have not been done within the last week, within 5 days after participant's last dose of study drug, the following tests and procedures will be performed:

* Participant will have a physical exam.
* Blood (about 3-4 tablespoons) and urine will be collected for routine tests. This blood will also be used to check participant's PSA levels, thyroid function, for biomarker testing, and to measure CTCs.
* Participant will have a bone scan and a CT or MRI scan of the chest, abdomen, pelvis, and any other area the study doctor thinks is needed to check the status of the disease.
* Participant will have a bone marrow aspiration and biopsy to check the status of the disease.
* Participant will fill out the questionnaire about pain.

Follow-Up Visit:

About 30 days after participant stops taking the study drug, the following procedures will be performed:

* Participant will have a physical exam.
* Blood (about 3-4 tablespoons) and urine will be collected for routine tests. This blood will also be used to check participant's PSA levels.

This is an investigational study. AMG208 is not FDA approved or commercially available. It is being used for research purposes only.

The study doctor can explain how the study drug is designed to work.

Up to 30 participants will be enrolled in this study. All will take part at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed adenocarcinoma of the prostate.
2. Presence of metastatic disease to the bone.
3. Patients must have a castrate level of testosterone (</= 50 ng/dL) at the screening visit, medical or surgically induced. For patients who are medically castrated, gonadotropin releasing hormone antagonist or analog must continue to maintain testicular suppression.
4. Evidence of progressive disease prior to enrolment based on AT LEAST one of the following criteria: a) Rising PSA: PSA progression defined by a minimum of two rising PSA levels with an interval of >/= 1 week between each determination. The PSA value at the Screening visit should be >/= 2 ng/mL; b) Non-measurable (evaluable) disease: 2 (two) or more new metastatic bone lesions by radionuclide bone scan or plain bone films (x-rays); c) Measurable disease (RECIST 1.1) by transaxial imaging: patients must show evidence of new or progressive disease on CT or MRI scans.
5. Eastern Cooperative Oncology Group (ECOG) performance status 0-2.
6. For patients who received combined androgen blockade (a GnRH antagonist, analog or orchiectomy in combination with continuous antiandrogen not including enzalutamide), disease progression must have been determined after antiandrogen discontinuation as defined below: a) For patients receiving flutamide: at least one of the PSA values must be obtained 4 weeks or more after flutamide discontinuation.; b) For patients receiving bicalutamide or nilutamide: at least one of the PSA values must be obtained 6 weeks or more after antiandrogen discontinuation.; However, in patients who did not respond to combined androgen blockade or who showed a decline in PSA for 3 months or less after an antiandrogen was administered as a second-line or later intervention, no withdrawal response will be expected and therefore disease progression will be determined provided at least one rising PSA value is obtained 2 weeks or more after antiandrogen discontinuation.
7. Patients who received any other hormonal therapy, including megestrol acetate, finasteride, ketoconazole, abiraterone, enzalutamide, diethylstilbestrol or any systemic corticosteroids, must have discontinued such agent for at least 2 weeks prior to enrollment. Progressive disease must be documented after discontinuation of such therapy. Low dose maintenance steroids (prednisone </=10 mg/d or hydrocortisone </= 30 mg/d equivalents) are permitted.
8. No more than two prior cytotoxic chemotherapies for metastatic prostate cancer.
9. Relative to Day 1 visit, at least 3 weeks since radiation therapy (2 weeks if single fraction), at least 4 weeks since major surgery or investigational therapy, and at least 8 weeks since radioisotope therapy.
10. Resolution of all acute toxic effects of prior therapy or surgical procedure to Grade </=1 at baseline.
11. Adequate organ function as defined: serum aspartate transaminase (AST) and serum alanine transaminase (ALT) </= 3 x upper limit of normal (ULN) if no metastatic liver involvement, or </= 5 if liver involvement; total serum bilirubin </= 1.5 x ULN; absolute neutrophil count (ANC) >/= 1500/uL; platelets >/= 100,000/uL; hemoglobin >/= 9.0 g/dL; serum albumin >/=3.0 g/dL; serum creatinine < 2.0 mg/dL or calculated creatinine clearance >/=60 ml/min; PT (or INR) or PTT </=1.5 x ULN. Subject may not have received any growth factors or blood transfusions within 7 days of the hematologic laboratory values obtained at the Screening visit.
12. Able to swallow the study drug and comply with study requirements.
13. Agree to use a double-barrier method of contraception, which involves the use of a condom in combination with one of the following: contraceptive sponge, diaphragm, or cervical ring with spermicidal gel or foam, if having sex with a woman of child-bearing potential during the length of the study and for at least one month after AMG 208 is discontinued.
14. Signed and dated informed consent document indicating that the patient (or legally acceptable representative) has been informed of all pertinent aspects of the trial prior to enrollment.

Exclusion Criteria:

1. Small cell or other variant histology.
2. Brain metastases or active epidural disease. Patients with treated epidural disease are eligible if stable for at least 4 weeks.
3. Diagnosis of any second malignancy within the last 2 years, except basal cell carcinoma, squamous cell skin cancer, or in situ carcinoma that has been adequately treated with no evidence of recurrent disease for 12 months.
4. Impending complication from bone metastasis (fracture and/or cord compression). Any bone fracture must be healed.
5. Presence of acute urinary obstruction.
6. Prior anti-c-Met or c-Met/VEGR-2 inhibitor.
7. Patients on stable doses of bisphosphonates or denosumab showing subsequent tumor progression may continue on this therapy; however, patients are not allowed to initiate bisphosphonate therapy in at least 4 weeks prior to or during the study.
8. Ongoing treatment with therapeutic doses (with therapeutic INR levels) of coumarin derivatives or oral anti-vitamin K agents. Therapeutic doses of low molecular weight heparins are allowed.
9. Concurrent or prior (within 14 days of study day 1) use of strong CYP3A4 inhibitors (including, but not limited to, ketoconazole, itraconazole, clarithromycin, indinavir, nefazodone, nelfinavir, ritonavir, saquinavir, telithromycin, voriconazole).
10. Concurrent or prior (within 7 days of study day 1) grapefruit products and other foods that are known to inhibit CYP3A4.
11. Concurrent or prior (within 28 days of study day 1) use of strong CYP3A4 inducers (including, but not limited to, dexamethasone, phenytoin, carbamazepine, rifampin, rifabutin, rifapentine, phenobarbital). Subjects should not take St John's Wort.
12. Concurrent or prior (within 28 days of study day 1) use of strong P-glycoprotein and Breast Cancer Receptor Protein inhibitors (including, but not limited to elacridar and valspodar).
13. Clinically significant cardiovascular disease including: a) Myocardial infarction within 6 months of Screening visit; b) Uncontrolled angina within 3 months of Screening visit; c) Current or past history of congestive heart failure NYHA class III or IV or history of anthracycline or anthracenedione (mitoxantrone) treatment, unless a screening echocardiogram or multi-gated acquisition scan (MUGA) performed within three months results in a left ventricular ejection fraction (LVEF) that is >/= 50%; d) History of clinically significant ventricular arrhythmias (e.g., ventricular tachycardia, ventricular fibrillation, torsade de pointes), grade >/= 2 cardiac dysrhythmias, atrial fibrillation of any grade, or QTcF interval > 470 msec on the screening Electrocardiogram (ECG); e) History of Mobitz II second degree or third degree heart block without a permanent pacemaker in place;
14. (Continued from Exclusion #13) f) Hypertension that cannot be controlled by medications (> 140 mmHg systolic OR > 90 diastolic despite optimal medical therapy).
15. Seizure disorder not controlled with standard medical therapy, or cerebrovascular accident or transient ischemic attack within 6 months of Screening visit.
16. Patients must not have clinical history of coagulopathy or bleeding diathesis, or arterial or venous thrombosis within 1 year of Screening visit.
17. Gastrointestinal abnormalities such as inability to take oral medication; requirement for intravenous alimentation; prior surgical procedures affecting absorption including total gastric resection; treatment for active peptic ulcer disease in the past 6 months; active gastrointestinal bleeding as evidenced by hematemesis, hematochezia or melena in the past 3 months without evidence of resolution documented by endoscopy or colonoscopy; malabsorption syndromes.
18. Other severe acute or chronic medical or psychiatric condition, or laboratory abnormality that would impart, in the judgment of the investigator, excess risk associated with study participation or study drugs administration, or which, in the judgment of the investigator would make the patient inappropriate for entry into the trial.
19. Current treatment on another therapeutic clinical trial.
20. Patients with known HIV, or active HBV or HCV infection
21. Concurrent medications that prolong QTc (e.g. levofloxacin, diphenhydramine, fluconazole) (Appendix F)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-10; Primary Completion 2019-10 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) | 6 weeks
  Progression free survival (PFS) defined as the time from treatment start to the time of clinical progression or death, whichever occurs first, or the time of last contact. The primary efficacy endpoint, PFS, continuously monitored using the Bayesian method by Thall et al.

CONTACTS AND LOCATIONS:
Overall Officials: Amado Zurita, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org